CLINICAL TRIAL: NCT02960919
Title: Prospective, Observational Study of Clinical Outcomes Among Children 2 to 59 Months of Age With Childhood Pneumonia and Other Co-morbidities in Lilongwe, Malawi Who Have Been Excluded From Pneumonia Clinical Trials
Brief Title: Innovative Treatments in Pneumonia (ITIP) 3
Status: Completed | Type: Observational
Sponsor: Save the Children (Other)
Collaborators: University of Washington (Other); University of North Carolina (Other); Kamuzu Central Hospital (Other); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: ITIP3
Record Dates: First submitted 2016-09-27; First posted 2016-11-10 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin; Penicillins; Gentamicins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oral amoxicillin or parenteral ampicillin/ penicillin and gentamicin
Drug: parenteral ampicillin/ penicillin
Drug: gentamicin

SUMMARY:
This is a prospective observational study assessing the clinical outcomes of children 2 to 59 months of age with both pneumonia and other co-morbidities presenting to a tertiary hospital outpatient setting in Malawi, Africa who are most at risk for mortality or have other complications and thus, are typically excluded from childhood pneumonia studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 2 to 59 months of age.
* Excluded from enrollment in Innovative Treatment in Pneumonia (ITIP) 1 and ITIP2 clinical trials due to presence of any of the following:
* Hypoxia (SaO2 < 90% on room air, as assessed by a pulse oximeter).
* Severe respiratory distress (e.g., presence of grunting, nasal flaring, head nodding, or severe chest-indrawing).
* Severe malaria, classified by World Health Organization (WHO) guidelines on hospital care for children, including a positive malaria rapid antibody test result.
* Severe anemia, classified by WHO Integrated Management of Childhood Illness (IMCI) guidelines (i.e., severe palmar pallor) only if a positive malaria rapid antibody test result.
* severe acute malnutrition (SAM) (i.e., weight for height/length < -3 SD, mid-upper arm circumference (MUAC) <115, or edema).
* HIV-1 seropositivity or HIV-1 exposure, assessed as follows: An HIV-positive result upon rapid antibody testing.
* If a child is less than 24 months of age and has an HIV-negative result upon rapid antibody test documented from the past three months, the child's biological mother's HIV status will need to be assessed. If the mother is HIV-positive, the child will be included. If the mother does not have documentation of an HIV-negative test result from the past 3 months, she will be tested via rapid antibody testing to determine the child's eligibility for this study.
* Ability and willingness of child's caregiver to provide informed consent and to be available for follow-up (in the inpatient ward, returning to KCH for a scheduled study follow-up visit, and by phone) for the planned duration of the study.

Exclusion Criteria:

* Possible tuberculosis (coughing for more than 14 days).
* Stridor when calm.
* Severe anemia, classified by WHO IMCI guidelines (i.e., severe palmar pallor) if a negative malaria rapid antibody test result.
* Known allergy to penicillin or amoxicillin.
* Receipt of an antibiotic treatment in the 48 hours prior to the study based on caregiver's self-report and/or documentation in child's medical record.
* Living outside Lilongwe urban area, the study catchment area.
* Any medical or psychosocial condition or circumstance that, in the opinion of the investigators, would interfere with the conduct of the study or for which study participation might jeopardize the child's health.
* Participation in a clinical study of an investigational product within 12 weeks prior to enrollment or planning to begin participation during this study.
* Prior participation in ITIP1, ITIP2 or ITIP3 during a previous pneumonia diagnosis.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 2 to 59 months of age who present to Kamuzu Central Hospital or Bwaila District Hospital with fast-breathing pneumonia or chest-indrawing pneumonia and other co-morbidities, or severe pneumonia AND are excluded from ITIP1 and ITIP2
Sampling Method: Non-Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes: cured, not cured | 14 days
  Clinically cured - absence of very fast-breathing, chest-indrawing, hypoxemia, severe respiratory distress (e.g., presence of grunting, nasal flaring, head nodding, or severe chest-indrawing), World Health Organization danger signs (i.e. lethargy or unconsciousness, convulsions, vomiting everything, or inability to drink or breastfeed), and fever:
  * Cured but failed initial antibiotic treatment regimen
  * Cured and did not fail initial antibiotic treatment regimen
  Not cured:
  * Deteriorating
  * Stable (not improving or deteriorating, prognosis unclear)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Ginsburg, MD MPH, Principal Investigator — Save the Children, Federation Inc
Locations (2):
- Malawi (2):
  - Bwaila District Hospital, Lilongwe
  - Kamuzu Central Hospital, Lilongwe

REFERENCES:
- [Derived] Mvalo T, McCollum ED, Fitzgerald E, Kamthunzi P, Schmicker RH, May S, Phiri M, Chirombo C, Phiri A, Ginsburg AS. Chest radiography in children aged 2-59 months enrolled in the Innovative Treatments in Pneumonia (ITIP) project in Lilongwe Malawi: a secondary analysis. BMC Pediatr. 2022 Jan 10;22(1):31. doi: 10.1186/s12887-021-03091-3. PMID 35012490
- [Derived] Ginsburg AS, Mvalo T, Hwang J, Phiri M, McCollum ED, Maliwichi M, Schmicker R, Phiri A, Lufesi N, May S. Malawian children with fast-breathing pneumonia with and without comorbidities. Pneumonia (Nathan). 2021 Feb 25;13(1):3. doi: 10.1186/s41479-021-00081-y. PMID 33627192